CLINICAL TRIAL: NCT03684902
Title: Burst Abdomen in Emergency Midline Laparotomy: Incidence and Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Maged, professor, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 43
Record Dates: First submitted 2018-09-24; First posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-09

CONDITIONS: Wound Dehiscence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- xpolration (Experimental): women who underwent emergency midline laprotomy
  Interventions: Procedure: emergency midline exploratory laparotomy

INTERVENTIONS:
Procedure: emergency midline exploratory laparotomy — Once an adequate level of anesthesia has been reached, the initial incision into the skin may be made. A scalpel is first used to cut into the superficial layers of the skin.with the diathermy The incision is then continued through the subcutaneous fat, the abdominal muscles, and finally, the peritoneum. (Morris J ;2017) For all the patients, closure of midline laparotomy wound was en-mass closure done with non-absorbable No. 1 (Polypropylene) or slowly absorbable (PDS) (double loop). sutures in continuous single layer fashion with 1 cm interval. (Morris J ;2017) The operative details were recorded with special consideration to the operative diagnosis, presence and types of adhesions, duration of surgery, the need for diversion and stoma formation, the use of intraperitoneal drain and the suture material to close the rectus sheath.
  Other Names: midline exploratory laparotomy

SUMMARY:
The study was conducted in 250 patients who underwent midline Laparotomy at Kasr Al-Ainy emergency department, Cairo University from August 2017 until March 2018. Factors such as age ,sex, body mass index, substance abuse, previous laparotomy, malignancy, diabetes mellitus , ascites, albumin, renal functions, bilirubin, hemoglobin, intra-abdominal pathology, suture material, creation of stoma, post-operative chest infection, , post-operative paralytic ileus, leakage and wound infection were observed and analyzed with odds ratio and P value

DETAILED DESCRIPTION:
General Anaesthesia can be appropriate for patients undergoing abdominal surgery. In common practice with rapid sequence induction with inhalational anesthetics (sevoflourane or isoflourane), opioids (fentanyl 1-2 mic/kg with induction & morphine 0.1 mg/kg) and neuromuscular blockers (succinylcholine 0.5 mg/kg or roucroinium 0.9 mg/kg) are used in general anesthesia for abdominal surgical procedures.

Once an adequate level of anesthesia has been reached, the initial incision into the skin may be made. A scalpel is first used to cut into the superficial layers of the skin.with the diathermy The incision is then continued through the subcutaneous fat, the abdominal muscles, and finally, the peritoneum.

For all the patients, closure of midline laparotomy wound was en-mass closure done with non-absorbable No. 1 (Polypropylene) or slowly absorbable (PDS) (double loop). sutures in continuous single layer fashion with 1 cm interval.

The operative details were recorded with special consideration to the operative diagnosis, presence and types of adhesions, duration of surgery, the need for diversion and stoma formation, the use of intraperitoneal drain and the suture material to close the rectus sheath.

During the postoperative period, VAS assessment of postoperative pain at 1 , and 24 hours, time of ambulation, time of oral feeding, hospital stay, and postoperative hemoglobin were recorded.Any postoperative complication especially chest infection, wound infection, postoperative leakage and postoperative paralytic ileus were reported.

Follow up of all cases was done weekly after discharge for 4 weeks. Examination of wound included inspection for any redness, edema or presence of discharge like pus or serosanguinous fluid. Special attention was given to maintain asepsis. Broad spectrum intravenous antibiotics The antibiotic therapy for the treatment of intra-abdominal infections greatly varies according to the infection severity. It is, in fact, possible to distinguish the intra-abdominal infections in three different categories. Mild infections should be treated promptly with surgical drainage and a short term therapy with a wide range antibiotic including anaerobes (ampicillin/sulbactam, cefoxitin). Mild-moderate infections which are largely the most frequent in the clinical practice should be also treated with a single drug which include anaerobes in its spectrum. Finally severe infections require a more aggressive therapeutic approach with a combination treatment covering anaerobes (clyndamicin, metronidazole), Gram negative rods (ciprofloxacin, aminoglycosides) and Gram positive cocci (penicillins, cephalosporins) including MRSA (glycopetides) and/or VRE (linezolid). with anaerobic coverage was started for all cases and later changed according to culture and sensitivity report.

During follow up duration, the participants were assigned to one of two groups. Group I involved patients developed burst abdomen whether partial (bowel not eviscerated) or complete (bowl not eviscerated) and group II involved those who didn't develop it. Half of Sutures were removed after 10 days , all the sutures removed after 14 days.

ELIGIBILITY:
Inclusion Criteria:

* All participants were subjected to emergency midline exploration.
* All participants at any age
* both sexes were included

Exclusion Criteria:

* those who arrested on table or at the immediate postoperative period

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2017-08-05 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
wound infection | 4 weeks after surgery
  redness, hotness, swelling of the wound

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed maged, MD, Principal Investigator — Professor
Locations (1):
- Kasr Alainy medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided